CLINICAL TRIAL: NCT00029380
Title: Sibling Donor Cord Blood Banking and Transplantation
Brief Title: Cord Blood Transplantation for Sickle Cell Anemia and Thalassemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Bertram H. Lubin, Children's Hospital, Oakland
Purpose: Treatment
Other Study IDs: 141; U01HL061877 (NIH)
Record Dates: First submitted 2002-01-10; First posted 2002-01-11 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-09

CONDITIONS: Hematologic Diseases; Anemia, Sickle Cell; Beta-Thalassemia; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Diseases; Anemia, Sickle Cell; beta-Thalassemia | interventions — Cyclophosphamide; Busulfan; Mycophenolic Acid; Cyclosporine; Cord Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: Sangstat
Drug: Cyclophosphamide
Drug: Busulfan
Drug: Mycophenolate Mofetil
Drug: Cyclosporine
Procedure: Cord Blood Transplantation

SUMMARY:
This study will develop a national cord blood bank for siblings of patients with hemoglobinopathies and thalassemia.

DETAILED DESCRIPTION:
BACKGROUND:

During the past decade, a number of advances have been made in the treatment of patients with sickle cell anemia and thalassemia. Among these advances is allogeneic bone marrow transplantation, which is the only current treatment that offers a potential for cure. In sickle cell anemia, transplantation has been performed in patients who have had advanced organ damage. In thalassemia, transplantation has been performed before having any evidence of iron-related tissue damage. Due to concerns over engraftment and graft versus host disease (GVHD), transplants for patients with hemoglobinopathies have been limited to situations in which a human leukocyte antigen (HLA) compatible donor existed. Unfortunately, an HLA-matched related donor is often not available. Umbilical cord blood (UCB), a recently recognized source of hematopoietic stem cells, has been used to successfully transplant bone marrow to over 500 patients. The potential advantage of cord blood over other donor sources of stem cells is the minimal risk of high-grade GVHD (even without complete HLA compatibility).

DESIGN NARRATIVE:

This study will establish a national sibling donor cord blood (SDCB) program, evaluate its use in a multi-center pilot study of transplantation, and develop a Web-based data management system to support these two projects. A multi-center pilot study was conducted on cord blood transplantation in children with either sickle cell disease or thalassemia. The investigators tested the hypothesis that a novel immunosuppressive conditioning regimen (fludarabine, cyclophosphamide, and busulfan) and post transplant therapy (mycophenolate mofetil and cyclosporine) would improve engraftment rates and prevent disease recurrence. The effect of SDCB transplantation on hematologic parameters and GVHD was monitored. Enrollment in the study was suspended on December 29, 2003. The protocol was revised, replacing the previous conditioning regimen of fludarabine, busulfan, and cyclophosphamide with a more conventional regimen of rabbit anti-thymocyte globulin (Sangstat), busulfan, and cyclophosphamide. The revised protocol is open for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Suitable UCB collection from an HLA-identical sibling
* Sickle cell anemia (Hb SS or S beta thalassemia) with significant disease manifestations as defined by at least one of the following criteria:

  1. A history of painful events defined as three or more painful events in the 2 years prior to enrollment. Pain may occur in typical sites associated with vaso-occlusive painful events and cannot be explained by causes other than sickle cell disease. The pain must last at least 4 hours and require treatment with either parenteral narcotics, an equianalgesic dose of oral narcotics (if pain is treated in a local facility where parenteral narcotics are not routinely used to treat painful events), or parenteral nonsteroidal anti-inflammatory drugs. Painful events managed at home will be considered only if there is documentation of the event in a clinical record that may be reviewed by an investigator.
  2. Acute chest syndrome (ACS) with two or more episodes of ACS with the development of a new infiltrate on chest radiograph and/or having a perfusion defect demonstrable on a lung radioisotope scan
  3. Any combination of painful events and episodes of ACS that total three events in the 2 years before transplantation
  4. Any clinically significant neurologic event (stroke or hemorrhage) or any neurologic defect lasting more than 24 hours
  5. Abnormal cerebral MRI and abnormal cerebral MRA
  6. An episode of dactylitis in the first year of life with significant anemia (Hbg less than 7 g/dL), or leukocytosis in the second year of life such that the risk of a severe adverse outcome before 18 years of age exceeds 54% (as defined by the cooperative study of sickle cell disease (CSSCD) infant cohort study)
  7. History of positive trans-cranial Doppler studies (average greater than 200 cm/sec)
* Beta thalassemia major with significant disease manifestations as defined by the following criteria: Beta thalassemia genotype consistent with clinical diagnosis of beta thalassemia major (could include patients with E-beta thalassemia genotype) and requiring eight or more red blood cell (RBC) transfusions a year and iron chelation therapy. Younger patients who are at risk of transfusional iron overload but who have not yet initiated iron chelation therapy will be eligible.
* Adequate physical function as measured by the following criteria:

  1. Cardiac: Asymptomatic or, if symptomatic, then left ventricular ejection fraction at rest must be greater than 40% and must improve with exercise, or shortening fraction greater than 26%
  2. Hepatic: Less than 5 times the clinical baseline of AST and less than 2.5 times the clinical baseline mg/dL of total serum bilirubin (clinical baseline is determined from the mean of the four most recent test results)
  3. Renal: Serum creatinine within normal range for age or if serum creatinine is outside normal range for age then renal function (creatinine clearance or GFR) greater than 50% of the lower limit of normal (LLN) for age
  4. Pulmonary: Asymptomatic, or, if symptomatic, DLCO, FEV1, FEC (diffusion capacity) greater than 45% of predicted (corrected for hemoglobin); if unable to obtain PFT, oxygen saturation greater than 85% on room air

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 1999-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Hematologic parameters
GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Victor Aquino, Study Chair — University of Texas Southwestern Medical Center - Dallas; Nancy Bunin, Study Chair — Children's Hospital of Philadelphia; Martin Champagne, Study Chair — Hopital Ste-Justine; Joel Brochstein, Study Chair — Hackensack Meridian Health; Michael Joyce, Study Chair — Nemours Children's Clinic; Naynesh Kamani, Study Chair — Children's National Research Institute; Gary Kleiner, Study Chair — University of Miami Batchelor Children's Research Center; Joanne Kurtzberg, Study Chair — Duke University Medical Center Children's Hospital; Bertram H. Lubin, Study Chair — UCSF Benioff Children's Hospital Oakland; Alexis Thompson, Study Chair — Ann & Robert H Lurie Children's Hospital of Chicago; Donna Wall, Study Chair — Texas Transplant Institute; Mark Walters, Study Chair — UCSF Benioff Children's Hospital Oakland; Lolie Yu, Study Chair — Louisiana State University Children's Medical Center
Locations (15):
- United States (14):
  - Children's Hospital Oakland, Oakland, California
  - Children's Hospital, Oakland, Oakland, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Batchelor Children's Research Center, Miami, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Louisiana State University Children's Medical Center, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University Medical Center Children's Hospital, Durham, North Carolina
  - Children's Hospital Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
- Hopital Ste-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Background] Reed W, Walters M, Lubin BH. Collection of sibling donor cord blood for children with thalassemia. J Pediatr Hematol Oncol. 2000 Nov-Dec;22(6):602-4. doi: 10.1097/00043426-200011000-00031. PMID 11132238
- [Background] Lubin BH, Eraklis M, Apicelli G. Umbilical cord blood banking. Adv Pediatr. 1999;46:383-408. No abstract available. PMID 10645470
- [Background] Woodard P, Lubin B, Walters CM. New approaches to hematopoietic cell transplantation for hematological diseases in children. Pediatr Clin North Am. 2002 Oct;49(5):989-1007. doi: 10.1016/s0031-3955(02)00026-3. PMID 12430622
- [Background] Reed W, Smith R, Dekovic F, Lee JY, Saba JD, Trachtenberg E, Epstein J, Haaz S, Walters MC, Lubin BH. Comprehensive banking of sibling donor cord blood for children with malignant and nonmalignant disease. Blood. 2003 Jan 1;101(1):351-7. doi: 10.1182/blood-2002-02-0394. Epub 2002 Aug 8. PMID 12393579
- [Background] Locatelli F, Rocha V, Reed W, Bernaudin F, Ertem M, Grafakos S, Brichard B, Li X, Nagler A, Giorgiani G, Haut PR, Brochstein JA, Nugent DJ, Blatt J, Woodard P, Kurtzberg J, Rubin CM, Miniero R, Lutz P, Raja T, Roberts I, Will AM, Yaniv I, Vermylen C, Tannoia N, Garnier F, Ionescu I, Walters MC, Lubin BH, Gluckman E; Eurocord Transplant Group. Related umbilical cord blood transplantation in patients with thalassemia and sickle cell disease. Blood. 2003 Mar 15;101(6):2137-43. doi: 10.1182/blood-2002-07-2090. Epub 2002 Nov 7. PMID 12424197
- [Background] Reed W, Walters M, Trachtenberg E, Smith R, Lubin BH. Sibling donor cord blood banking for children with sickle cell disease. Pediatr Pathol Mol Med. 2001 Mar-Apr;20(2):167-74. PMID 12673840
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296